CLINICAL TRIAL: NCT01907581
Title: Impact of Socio-economic Vulnerability on Initial Severity and Prognosis in Patients Admitted to an ICU. Prospective, Multi-centre Cohort Study
Brief Title: Impact of Socio-economic Vulnerability on Initial Severity and Prognosis in Patients Admitted to an ICU.
Acronym: IVOIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Quenot PHRC IR 2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Patients at Intensive Care Unit

ARMS (1):
- Patients admitted to an ICU (Other)
  Interventions: Other: Quality of life questionnaires

INTERVENTIONS:
Other: Quality of life questionnaires

SUMMARY:
A gravity admission largest resuscitation and a poorer prognosis are expected for patients experiencing socio-economic vulnerability. This is the first study in France and investigating the field of resuscitation which will allow us to have a vision of the French health system and its consequences. The frequency of PTSD is expected to be more important in this vulnerable population itself with quality of life at discharge worse. The results of this study are a prerequisite for the implementation of preventive measures targeted and more suitable for those patients experiencing socio-economic vulnerability remediation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have been informed about the study (directly or via a person of trust) and have given their consent
* Patients admitted to intensive care in accordance with the criteria defined by decree n° 2002-465 of the law of 05th April 2002 relative to the rights of patients and the quality of the healthcare system. It concerns patients who present or are likely to present life-threatening acute multi-organ failure requiring support care involving at least one of the following procedures: invasive or non-invasive mechanical ventilation, continuous or discontinuous hemofiltration, dobutamine, adrenaline, noradrenaline, ECMO

Exclusion Criteria:

* - Refusal to take part,
* Age < 18 years
* Adult under guardianship (or ward of court),
* Patients impossible to follow for 3 months (concomitant disease not related to the admission to the ICU that may cause death within 3 months….),
* Patients presenting major cognitive impairment that precludes a reliable interview,
* Patients and/or close relatives/friends who cannot be questioned or cannot provide information,
* Absence of a family and/or close friends

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1417 (Actual)
Dates: Start 2013-06-08 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Severity at admission assessed by the SAPS II score at ICU admission | Within the first 24 hours of hospitalization in intensive care
Rate of mortality within 3 months following ICU admission | within 3 months following ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Result] Quenot JP, Helms J, Labro G, Dargent A, Meunier-Beillard N, Ksiazek E, Bollaert PE, Louis G, Large A, Andreu P, Bein C, Rigaud JP, Perez P, Clere-Jehl R, Merdji H, Devilliers H, Binquet C, Meziani F, Fournel I; IVOIRE Trial Investigators and the CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). Influence of deprivation on initial severity and prognosis of patients admitted to the ICU: the prospective, multicentre, observational IVOIRE cohort study. Ann Intensive Care. 2020 Feb 11;10(1):20. doi: 10.1186/s13613-020-0637-1. PMID 32048075